CLINICAL TRIAL: NCT01003405
Title: A Open-label, Long-term Extension Study of KUC-7483 in Patients With Overactive Bladder
Brief Title: Long-term Safety and Efficacy of KUC-7483 in Patients With Overactive Bladder
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUC1302
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Frequency; Micturition; Urgency; Urge urinary incontinence; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — ritobegron ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KUC-7483 (Experimental)
  Interventions: Drug: KUC-7483

INTERVENTIONS:
Drug: KUC-7483

SUMMARY:
To investigate the long-term safety, efficacy and pharmacokinetics of KUC-7483 in patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed the Phase III double-blind study.

Exclusion Criteria:

* Patients with serious adverse events or clinically significant adverse events in the Phase III double-blind study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
The long-term safety of KUC-7483 for the treatment of overactive bladder. | 52 weeks

SECONDARY OUTCOMES:
The long-term efficacy of KUC-7483 for the treatment of overactive bladder. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Clinical Development Department, Kissei pharmaceutical Co., Ltd.
Locations (1):
- Japan, Hokkaido,Tohoku,Kanto,Chubu,Kansai,Shikoku,Kyushu, Japan